CLINICAL TRIAL: NCT02393560
Title: A Study to Determine the Presence and Volume of Monosodium Urate Crystals as Assessed by Dual-Energy Computed Tomography in Gout Patients Treated With Allopurinol
Brief Title: DECT Study in Allopurinol-Treated Gout Patients
Status: Completed | Type: Observational
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALLO-402
Record Dates: First submitted 2015-03-15; First posted 2015-03-19 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood sample may be used for optional genetic testing in subjects who give consent. Serum aliquots will be collected and may be used for the analysis of potential analytes and biomarkers, but may not be used for genetic testing without the subject's written consent.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gout subjects on stable dose of allopurinol (at least 300mg)
  Interventions: Procedure: DECT scan

INTERVENTIONS:
Procedure: DECT scan

SUMMARY:
The purpose of this study is to determine presence and volume of monosodium urate (MSU) crystal deposits as determined by dual-energy computed tomography (DECT) imaging in gout subjects treated with allopurinol with and without visible tophi.

DETAILED DESCRIPTION:
DECT is a technique that enables visualization of MSU crystal deposits by analysis of the chemical composition of the scanned materials. This study will determine the extent of MSU crystal volume in the hands/wrists, feet/ankles, and knees as determined by DECT of subjects with gout taking a dose of at least 300 mg allopurinol daily for the past 12 weeks.

Patients with gout on allopurinol with and without tophi to be assessed using DECT imaging for crystal deposition with assessments, which include patient and provider assessments of disease severity and pain, prior to and after the scan.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the study procedures, the risks involved and willing to provide written informed consent before the first study related activity.
* Subject is willing to adhere to the visit/protocol schedules.
* Subject meets the diagnosis of gout as per the American Rheumatism Association Criteria for the Classification of Acute Arthritis of Primary Gout.
* Subject has been taking allopurinol at a dose of at least 300 mg daily for at least 12 weeks prior to Day 1, as the sole uratelowering therapy.

Exclusion Criteria:

* Subject who is pregnant or breastfeeding.
* Subject with any other medical or psychological condition, which in the opinion of the Investigator and/or Medical Monitor, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements (including dual energy computed tomography imaging), or to complete the study.
* Subject who has received an investigational therapy or has participated in any clinical trial or research study within 30 days of Day 1.
* Subject who has taken pegloticase (KRYSTEXXA®) or is expected to take pegloticase during the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gout subjects taking a stable dose of at least 300 mg allopurinol daily for at least 12 weeks prior to Day 1 as the sole urate-lowering therapy
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Presence and volume of MSU crystal deposits as determined by DECT imaging | 8 weeks

SECONDARY OUTCOMES:
Joint erosion as visualized on DECT images | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nihar Bhakta, MD, Study Director — Ardea Biosciences, Inc.
Locations (10):
- United States (9):
  - Irvine, California
  - Englewood, Colorado
  - Wheat Ridge, Colorado
  - Atlanta, Georgia
  - Cleveland, Ohio
  - Lyndhurst, Ohio
  - Willoughby Hills, Ohio
  - Dallas, Texas
  - Plano, Texas
- Grafton, Auckland, New Zealand